CLINICAL TRIAL: NCT07392424
Title: BreastCancerPEP: A Randomized Trial of a Six-Month Online Empowerment Program to Improve Mental and Physical Health in Women With Breast Cancer
Brief Title: BreastCancerPEP: A Six-Month Online Empowerment Program to Improve Mental and Physical Health in Women With Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gabriela Ilie (Other)
Collaborators: Nova Scotia Health Authority (Other); Dalhousie University (Other); Queen Elizabeth II Health Sciences Centre (Other)
Responsible Party: Sponsor-Investigator, Gabriela Ilie, Associate Professor, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: BreastCancerPEP-RCT-2026
Record Dates: First submitted 2025-11-21; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: empowerment; mental health; patient activation; health promotion; breast cancer; quality of life; psychological distress; digital health; self-management; patient-reported outcomes; patient-centred care; lifestyle intervention; cancer survivorship
MeSH Terms: conditions — Breast Neoplasms; Empowerment; Psychological Well-Being; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Intervention (Experimental) (Experimental): Participants randomized to the Early Intervention arm will begin the Breast Cancer Patient Empowerment Program (Breast Cancer PEP) immediately after baseline assessment. The 6-month, home-based digital program includes daily emails with structured physical activity guidance, arm and shoulder rehabilitation exercises, mindfulness practices, and lifestyle education modules, along with optional peer-support check-ins and monthly videoconference sessions. Participants complete weekly self-report compliance surveys throughout the 6-month program.
  Interventions: Behavioral: Breast Cancer Patient Empowerment Program (BreastCancerPEP)
- Delayed Intervention / Wait-List Control (Active Comparator) (Active Comparator): Participants randomized to the Delayed Intervention arm receive usual care for the first 6 months following baseline assessment. No program materials or intervention content are provided during this period. At approximately 6 months, participants complete follow-up assessments and then begin the same 6-month Breast Cancer Patient Empowerment Program (Breast Cancer PEP) as the Early Intervention arm, including daily digital content, rehabilitation exercises, mindfulness practices, lifestyle modules, optional peer-support, and monthly videoconference sessions.
  Interventions: Behavioral: Breast Cancer Patient Empowerment Program (BreastCancerPEP)

INTERVENTIONS:
Behavioral: Breast Cancer Patient Empowerment Program (BreastCancerPEP) — The Breast Cancer Patient Empowerment Program (Breast Cancer PEP) is a 6-month, home-based digital behavioural intervention delivered through daily automated emails containing structured physical activity guidance, resistance-band and body-weight strength training, yoga and stretching routines, arm and shoulder rehabilitation exercises, mindfulness and relaxation practices, and lifestyle education modules. Optional peer-support check-ins and monthly videoconference group sessions are included. Intervention content is standardized through a 182-day pre-programmed email and video library. Participants in both study arms receive the same intervention content, with timing dependent on randomization assignment.

SUMMARY:
This study is evaluating a six-month, home-based Patient Empowerment Program (Breast Cancer PEP) for women receiving treatment for newly diagnosed invasive breast cancer. The program provides daily guidance on physical activity, arm and shoulder rehabilitation, stress-reduction practices, healthy lifestyle habits, and social support, all delivered through online videos, emails, and optional group sessions.

The purpose of the study is to learn whether this program can reduce psychological distress and improve overall well-being compared with standard cancer care. Psychological distress will be measured using a simple questionnaire called the Kessler Psychological Distress Scale (K10). The study will also look at general health, quality of life, and participants' experiences with the program.

A total of 160 women across Nova Scotia will take part. Participants will be randomly assigned to start the program right away or to receive standard care for six months before getting access to the program. Everyone will complete online questionnaires at the beginning of the study and again at 6 and 12 months. A small number of participants may also be invited to take part in optional interviews to share their experiences.

Researchers will also explore how participants use the digital program, what parts are most helpful, and whether the program could be offered more broadly in the future. The trial is being conducted across all Nova Scotia Health zones and coordinated through the QEII Health Sciences Centre.

DETAILED DESCRIPTION:
Breast Cancer PEP (BC-PEP) is a six-month, home-based, digitally delivered supportive-care program designed for individuals undergoing treatment for newly diagnosed invasive breast cancer. The program integrates physical activity, upper-limb rehabilitation, mindfulness, nutrition education, and self-management strategies. BC-PEP is based on prior PEP programs evaluated in Atlantic Canada, which demonstrated high feasibility and strong participant engagement.

In this randomized, wait-list-controlled trial, participants assigned to the early-intervention arm begin the 6-month BC-PEP program immediately after randomization, while participants in the wait-list control arm receive standard care for 6 months before initiating the same program. All participants are followed for approximately 12 months to assess intervention effects and longer-term outcomes. Randomization and allocation procedures are conducted centrally, and the study is implemented across multiple Nova Scotia Health sites.

Intervention Delivery:

BC-PEP is delivered primarily through automated daily emails generated via REDCap over 182 consecutive days. Each email provides a structured set of activities, including:

Progressive aerobic activity designed to meet oncology-specific guidelines Twice-weekly resistance-training sessions using household equipment or elastic bands Daily stretching and upper-limb rehabilitation exercises aligned with surgical recovery timelines A 10-minute daily mindfulness or relaxation practice Short educational modules addressing sleep, stress coping, communication, body image, and nutrition

Participants have access to a video library with instructional content, may engage in an optional peer-support "buddy system," and are invited to monthly videoconference sessions with study clinicians.

Implementation and Engagement Monitoring Engagement metrics are collected throughout the program, including weekly adherence surveys, email-open rates, video-view data, and participation in monthly sessions. Implementation outcomes will be examined using a Hybrid Type I effectiveness-implementation approach guided by the RE-AIM framework.

This digital, low-cost program is designed to be scalable and accessible across diverse geographic regions. Study findings are intended to inform the effectiveness and implementation potential of BC-PEP as part of routine supportive cancer care.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria:

1. Age ≥ 18 years.
2. Diagnosis: Biopsy-confirmed invasive breast cancer.
3. Treatment Plan: Scheduled to undergo breast cancer surgery, with or without neoadjuvant chemotherapy.
4. Medical Safety for Exercise: Able to safely participate in low-to-moderate physical activity and light resistance training based on study screening. Participants with a history of myocardial infarction, stroke, or other significant cardiovascular conditions within the last 12 months require documented medical clearance from a Family Physician, Oncologist, or Cardiologist.
5. Residence: Resides in Nova Scotia and able to participate in a province-wide, digitally delivered program.
6. Digital Access and Literacy: Regular access to email and the internet on a computer, tablet, or smart phone. Able to open emailed links and navigate online videos and surveys (caregiver assistance permitted). Has an active email account or willingness to create one and check it daily.
7. Language Ability: Able to read, speak, and understand English sufficiently to follow program content and complete study questionnaires.
8. Study Participation Requirements: Willing and able to complete online questionnaires at baseline, 6 months, and 12 months. Willing to complete weekly self-reported compliance surveys during the 6-month intervention period.

Exclusion Criteria

Participants will be excluded if any of the following apply:

1. Medical Contraindications: Myocardial infarction, stroke, or other major cardiovascular event within the past 12 months without medical clearance indicating safety for exercise. Any medical, orthopedic, neurological, or other condition that would preclude safe participation in a home-based physical activity program.
2. Digital Access Limitations: Inability to access the internet or lack of a device necessary to receive daily emails or view program videos. Inability to navigate online videos or survey links, even with caregiver assistance.
3. Participation Limitations: Unwillingness or inability to complete required questionnaires or engage with digitally delivered program components.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2028-03-15 (Estimated); Study Completion 2029-03-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with clinically significant psychological distress (Kessler Psychological Distress Scale-10 ≥20) | 6 months after randomization (Day 183 ± 2 days)
  Proportion of participants scoring ≥20 on the Kessler Psychological Distress Scale-10 (K10) at 6 months after randomization. The K10 is a validated 10-item measure of psychological distress with scores ranging from 10-50, where higher scores indicate worse distress.

SECONDARY OUTCOMES:
Change in psychological distress (Kessler Psychological Distress Scale-10 total score) | Baseline to 6 months; baseline to 12 months
  Change in total score on the Kessler Psychological Distress Scale-10 (K10) from baseline to 6 and 12 months. The K10 ranges from 10-50, with higher scores indicating worse distress. This outcome complements the primary binary measure by assessing psychological distress as a continuous variable.
Change in health-related quality of life (SF-12v2 Physical and Mental Component Scores) | Baseline to 6 months; baseline to 12 months
  Change in SF-12v2 Physical Component Summary (PCS) and Mental Component Summary (MCS) scores from baseline to 6 and 12 months. Scores range from 0-100, with higher scores indicating better health status.
Change in health utility score (SF-6D) | Baseline to 6 months; baseline to 12 months
  Change in SF-6D health utility score derived from SF-12v2 responses. Scores range from approximately 0.29-1.00, with higher scores indicating better health-related quality of life.
Change in cancer-specific quality of life (EORTC QLQ-C30) | Baseline to 6 months; Baseline to 12 months.
  Change in EORTC QLQ-C30 domain scores. All scales transformed to 0-100. Higher scores indicate better functioning for functional scales and worse symptoms for symptom scales; higher global health = better QoL.
Change in breast cancer-specific quality of life (EORTC QLQ-BR23) | Baseline to 6 months; Baseline to 12 months.
  Change in QLQ-BR23 domain scores (0-100). Higher functional scores indicate better functioning; higher symptom scores indicate worse symptoms.
Change in self-efficacy (Self-Efficacy for Managing Chronic Disease 6-item Scale) | Baseline to 6 months; baseline to 12 months
  Change in SEMCD-6 total score. Scores range 1-10; higher scores indicate greater self-efficacy.
Change in patient activation (Patient Activation Measure-13) | Baseline to 6 months; baseline to 12 months
  Change in PAM-13 total score. Scores range 0-100; higher scores indicate greater activation.
Change in generalized anxiety symptoms (GAD-7) | Baseline to 6 months; baseline to 12 months
  Change in GAD-7 total score. Scores range 0-21; higher scores indicate greater anxiety.
  Time Frame: Baseline to 6 months; Baseline to 12 months.
Change in cognitive function (PROMIS® Short Form v2.0 - Cognitive Function 8a) | Baseline to 6 months; baseline to 12 months
  Change in PROMIS Cognitive Function 8a T-score. T-scores typically range ~20-80; higher T-scores indicate better cognitive function.
Change in upper-limb disability and symptoms (QuickDASH) | Baseline to 6 months; baseline to 12 months
  Change in QuickDASH total score. Scores range 0-100; higher scores indicate greater disability/symptoms (worse function).
Change in menopause symptoms (Menopause Quick 6) | Baseline to 6 months; baseline to 12 months
  Change in MQ-6 total score (6 items; scale scoring varies by version). Higher scores indicate more severe menopause symptoms.
Change in social support (Medical Outcomes Study Social Support Survey) | Baseline to 6 months; baseline to 12 months
  Change in MOS-SSS summary score (and/or subscales). Scores transformed to 0-100; higher scores indicate greater perceived social support.
Change in body weight (self-reported kilograms) | Baseline to 6 months; baseline to 12 months
  Change in participant self-reported body weight (kg) from baseline to 6 and 12 months.
Change in diet quality (Rapid Eating Assessment for Participants - Shortened v2) | Baseline to 6 months; baseline to 12 months
  Change in REAP-S v2 total score. Scores range from 0-60; higher scores indicate healthier dietary habits.
Self-reported adherence to cancer treatment | Baseline to 6 months; baseline to 12 months
  Proportion of participants reporting full adherence to prescribed cancer treatment(s) via questionnaire.
Clinically verified adherence to cancer treatment | Baseline to 6 months; baseline to 12 months
  Proportion of participants documented as adherent in medical records.
Number of hospitalizations (administrative data) | Baseline to 6 months; baseline to 12 months
  Count of all-cause hospitalizations per participant from linked administrative data.
Number of physician billing events (administrative data) | Baseline to 6 months; baseline to 12 months
  Count of physician billing events per participant from linked provincial administrative databases.

OTHER OUTCOMES:
Participant satisfaction with program components (0-10 rating scale) | At 6 months (post-intervention)
  Participant-reported satisfaction with individual components of the Breast Cancer PEP program, assessed via a post-intervention survey. Each component (e.g., aerobic exercise, diet, mindfulness practices) is rated on a 0-10 Likert-type scale, where 0 = not at all helpful and 10 = extremely helpful.
Participant adherence to program activities (weekly self-report surveys) | Throughout 6-month intervention
  Percentage of prescribed weekly PEP activities completed, based on participant self-report surveys.
Change in physical activity (self-reported minutes per week) | Baseline to 6 months; baseline to 12 months
  Change in self-reported weekly minutes of moderate-to-vigorous physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No